CLINICAL TRIAL: NCT02916316
Title: Prospective Observational Study Investigating the Cardiotoxicity of Anthracyclines in Patients With Diffuse Large B-Cell
Brief Title: Study Investigating the Cardiotoxicity of Anthracyclines in Patients With Diffuse Large B-Cell
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_Cardio-DLBCL
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Lymphoma; Large B-Cell; Diffuse Large B-Cell
Keywords: Lymphoma; Large B-Cell; Cardiotoxicity
MeSH Terms: conditions — Lymphoma; Cardiotoxicity | interventions — Doxorubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chemo immunotherapy: All patients enrolled in the study will have to be treated with a chemo immunotherapy scheme R-CHOP with doxorubicin, with doxorubicin analogue or non pegylated liposomal anthracycline (R-COMP; Sec. 648 DM) administered every 21 days for 6 cycles. In unfavourable patients (stage II-IV) are allowed 2 additional cycles of rituximab at the end of the 6 cycles of R-CHOP.
  Interventions: Drug: R-CHOP with doxorubicin

INTERVENTIONS:
Drug: R-CHOP with doxorubicin — Chemoimmunotherapy every 21 days for 6 cycles. In unfavourable patients (stage II-IV) are allowed 2 additional cycles of rituximab at the end of the 6 cycles of R-CHOP.
  Other Names: R-CHOP with doxorubicin analogue; R-COMP

SUMMARY:
All patients enrolled in the study will have to be treated with a chemo immunotherapy scheme R-CHOP with doxorubicin, with doxorubicin analogue or non pegylated liposomal anthracycline (R-COMP; Sec. 648 DM) administered every 21 days for 6 cycles. In unfavourable patients (stage II-IV) are allowed 2 additional cycles of rituximab at the end of the 6 cycles of R-CHOP.

DETAILED DESCRIPTION:
The study was designed as a prospective observational multicenter study to evaluate the role of possible early markers of cardiotoxicity estimating an overall maximum risk equal to 20% of patients. The sample size, required to obtain an estimate of conventional anthracycline cardiotoxicity in the population, has been calculated with a confidence interval of 95% and a maximum acceptable error of ± 0.075. According to the conditions described above, the sample size of patients treated with conventional anthracycline results to be 124 patients.

Considering a 10-15% of not evaluable patients, the sample size is fixed at 150 patients treated with R-CHOP. The duration of the enrollment phase is defined in 2 years.

With this sample size should be possible to assess the risk of cardiotoxicity related to predictors with a worst group frequency at least of 10%.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Diffuse Large B-Cell Lymphoma diagnosis
* Patient eligible to receive 6 cycles of R-CHOP or R-CHOP like chemotherapy at full doses
* Age ≥ 18
* Stage I-IV
* Written informed consent
* ECOG Performance Status 0-3
* Ventricular Ejection Fraction (VEF) ≥40%
* No previous treatment for lymphoma (except for RT-IF)
* Negative β-HCG pregnancy test result at diagnosis for female of childbearing potential
* Use of acceptable method of contraception during the study and for 3 months after receiving the last dose of study drug for patients with childbearing potential
* Availability of the patient to be followed for all the phases of the chemotherapy treatment and for the subsequent follow-up

Exclusion Criteria:

* Inability to schedule a treatment at full doses of chemoimmunotherapy R-CHOP or R-CHOP-like for different reasons
* Central nervous system involvement due to lymphoma
* HIV
* Active cardiac pathology including heart failure, left ventricular dysfunction documented by a LVEF <40%, arrhythmias (rapid atrial fibrillation, frequent ventricular arrhythmias), valvular aortic or mitral disfunction > moderate, ischemic heart disease (myocardial infarction or acute coronary syndrome for over 6 months, angina at rest or with mild efforts)
* Previous treatment for lymphoma
* Other malignancy in the 3 years prior to the diagnosis of lymphoma with exception of non-melanoma skin cancer or in situ carcinoma
* Any other co-existing medical condition that would preclude participation in the study (uncontrolled bacterial or viral or fungal infection)
* Pregnant, or lactating and breastfeeding female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diffuse Large B-Cell Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2014-02-12 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiotoxicity | 1 year from enrollment
  defined as the rate of cardiovascular events classified according to the Lenihan criteria 2013

SECONDARY OUTCOMES:
Overall response rate (ORR) | 6 months from enrollment
  defined according to international criteria (Cheson 2007)
Rate of response to treatment | 6 months from enrollment
  defined according to international criteria (Cheson 2007)
Overall survival (OS) | 3 years from enrollment
  It will be calculated for all patients enrolled in the study from the date of start of therapy to the date of death or last follow-up.
Progression-free survival (PFS) | 3 years from enrollment
  It will be calculated for all patients from the start of therapy given to the date of progression or death or last follow-up.
failure-free survival (FFS) | 3 years from enrollment
  It will be calculated for all patients from the therapy start date to the date of an event or last follow-up.
  The events considered for the FFS definition are the following: treatment discontinuation for toxicity, response <RC, relapse / progression, death for any cause.
Freedom From cardiovascular Event (FFCE) | 3 years from enrollment
  calculated for all patients from the therapy start date to the time of occurrence of a cardiovascular event as defined by primary endopoint or follow-up date.
Number of events recorded during the treatment and codified according to NCI-CTC v4.03 | 3 years from enrollment
  it will be defined by the number of events recorded during the treatment and codified according to NCI-CTC v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Guido Gini, MD, Principal Investigator — AOU Ospedali Riuniti, Ematologia ANCONA
Locations (18):
- Italy (18):
  - AO Riuniti Papardo Piemonte, Messina, ME
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Nuovo Ospedale Di Sassuolo S.P.A., Sassuolo, Modena
  - A.O. Universitaria Policlinico Di Modena, Modena, MO
  - Ospedali Riuniti Villa Sofia - Cervello, Palermo, PA
  - UO Ematologia e CTMO di Piacenza, Piacenza, PC
  - A.O. Universitaria Ospedali Riuniti - Ospedale Umberto I Di Ancona, Ancona
  - Ospedale S. Giacomo di Castelfranco Veneto, Castelfranco Veneto
  - Ospedale Riuniti di Foggia, Foggia
  - UO Ematologia PO Vito Fazzi, Lecce
  - AOU Universitа degli Studi della Campania Luigi Vanvitelli, Napoli
  - Istituto Oncologico Veneto, Padua
  - U.O. Complessa di Ematologia Ospedale di Parma, Parma
  - Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ematologia e Trapianto Istituto Regina Elena IFO, Roma
  - Osp.Sant'Eugenio Divisione di Ematologia, Roma
  - Ospedale Ca Foncello, Treviso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris NL, Jaffe ES, Stein H, Banks PM, Chan JK, Cleary ML, Delsol G, De Wolf-Peeters C, Falini B, Gatter KC, et al. A revised European-American classification of lymphoid neoplasms: a proposal from the International Lymphoma Study Group. Blood. 1994 Sep 1;84(5):1361-92. No abstract available. PMID 8068936
- [Background] Fisher RI, Gaynor ER, Dahlberg S, Oken MM, Grogan TM, Mize EM, Glick JH, Coltman CA Jr, Miller TP. Comparison of a standard regimen (CHOP) with three intensive chemotherapy regimens for advanced non-Hodgkin's lymphoma. N Engl J Med. 1993 Apr 8;328(14):1002-6. doi: 10.1056/NEJM199304083281404. PMID 7680764
- [Background] International Non-Hodgkin's Lymphoma Prognostic Factors Project. A predictive model for aggressive non-Hodgkin's lymphoma. N Engl J Med. 1993 Sep 30;329(14):987-94. doi: 10.1056/NEJM199309303291402. PMID 8141877
- [Background] Tilly H, Lepage E, Coiffier B, Blanc M, Herbrecht R, Bosly A, Attal M, Fillet G, Guettier C, Molina TJ, Gisselbrecht C, Reyes F; Groupe d'Etude des Lymphomes de l'Adulte. Intensive conventional chemotherapy (ACVBP regimen) compared with standard CHOP for poor-prognosis aggressive non-Hodgkin lymphoma. Blood. 2003 Dec 15;102(13):4284-9. doi: 10.1182/blood-2003-02-0542. Epub 2003 Aug 14. PMID 12920037
- [Background] Pfreundschuh M, Trumper L, Kloess M, Schmits R, Feller AC, Rudolph C, Reiser M, Hossfeld DK, Metzner B, Hasenclever D, Schmitz N, Glass B, Rube C, Loeffler M; German High-Grade Non-Hodgkin's Lymphoma Study Group. Two-weekly or 3-weekly CHOP chemotherapy with or without etoposide for the treatment of young patients with good-prognosis (normal LDH) aggressive lymphomas: results of the NHL-B1 trial of the DSHNHL. Blood. 2004 Aug 1;104(3):626-33. doi: 10.1182/blood-2003-06-2094. Epub 2004 Feb 24. PMID 14982884
- [Background] Pfreundschuh M, Trumper L, Kloess M, Schmits R, Feller AC, Rube C, Rudolph C, Reiser M, Hossfeld DK, Eimermacher H, Hasenclever D, Schmitz N, Loeffler M; German High-Grade Non-Hodgkin's Lymphoma Study Group. Two-weekly or 3-weekly CHOP chemotherapy with or without etoposide for the treatment of elderly patients with aggressive lymphomas: results of the NHL-B2 trial of the DSHNHL. Blood. 2004 Aug 1;104(3):634-41. doi: 10.1182/blood-2003-06-2095. Epub 2004 Mar 11. PMID 15016643
- [Background] Balzarotti M, Spina M, Sarina B, Magagnoli M, Castagna L, Milan I, Ripa C, Latteri F, Bernardi D, Bertuzzi A, Nozza A, Roncalli M, Morenghi E, Tirelli U, Santoro A. Intensified CHOP regimen in aggressive lymphomas: maximal dose intensity and dose density of doxorubicin and cyclophosphamide. Ann Oncol. 2002 Sep;13(9):1341-6. doi: 10.1093/annonc/mdf242. PMID 12196358
- [Background] Vitolo U, Liberati AM, Cabras MG, Federico M, Angelucci E, Baldini L, Boccomini C, Brugiatelli M, Calvi R, Ciccone G, Genua A, Deliliers GL, Levis A, Parvis G, Pavone E, Salvi F, Sborgia M, Gallo E; Intergruppo Italiano Linfomi. High dose sequential chemotherapy with autologous transplantation versus dose-dense chemotherapy MegaCEOP as first line treatment in poor-prognosis diffuse large cell lymphoma: an "Intergruppo Italiano Linfomi" randomized trial. Haematologica. 2005 Jun;90(6):793-801. PMID 15951292
- [Background] Wilson WH. Chemotherapy sensitization by rituximab: experimental and clinical evidence. Semin Oncol. 2000 Dec;27(6 Suppl 12):30-6. PMID 11225998
- [Background] Demidem A, Lam T, Alas S, Hariharan K, Hanna N, Bonavida B. Chimeric anti-CD20 (IDEC-C2B8) monoclonal antibody sensitizes a B cell lymphoma cell line to cell killing by cytotoxic drugs. Cancer Biother Radiopharm. 1997 Jun;12(3):177-86. doi: 10.1089/cbr.1997.12.177. PMID 10851464